CLINICAL TRIAL: NCT00641719
Title: A Superiority Study of LY248686 Versus Placebo in the Treatment of Patients With Diabetic Peripheral Neuropathic Pain - Extension Phase
Brief Title: A Long-term Study for the Treatment of Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12194; F1J-JE-HMFY (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Results first posted 2011-03-31 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duloxetine 40 mg (Experimental): Duloxetine 40 milligrams (mg) once daily (QD), orally (PO), 1 year
  Interventions: Drug: Duloxetine hydrochloride
- Duloxetine 60 mg (Experimental): Duloxetine 60 mg QD, PO, 1 year
  Interventions: Drug: Duloxetine hydrochloride

INTERVENTIONS:
Drug: Duloxetine hydrochloride — Duloxetine 40 mg QD, PO, 1 year
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 40 mg
Drug: Duloxetine hydrochloride — Duloxetine 60 mg QD, PO, 1 year
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine 60 mg

SUMMARY:
The purpose of the study is to investigate safety and efficacy of duloxetine for patients with painful diabetic neuropathy at long-term use.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have completed the 13-week treatment in the preceding study (Protocol No. 0715N0831: NCT00552175).
* Patients who desire to receive continued treatment with LY248686 from the preceding study.
* Patients with latest glycosylated hemoglobin (HbA1c) ≤9.0% before Visit 7.
* Patients who can provide written consent in person.

Exclusion Criteria:

* Patients who concurrently have serious cardiovascular, hepatic, renal, respiratory, or blood disease, or symptomatic peripheral vascular disease, and thus are considered inappropriate to be included in the study.
* Pregnant patients or women who desire to become pregnant during the study period, and breast feeding patients.
* Other patients judged by the investigator/subinvestigator to be inappropriate as a subject in this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- Japan (25):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aomori
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gunma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ibaraki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokushima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama

REFERENCES:
- [Derived] Yasuda H, Hotta N, Kasuga M, Kashiwagi A, Kawamori R, Yamada T, Baba Y, Alev L, Nakajo K. Efficacy and safety of 40 mg or 60 mg duloxetine in Japanese adults with diabetic neuropathic pain: Results from a randomized, 52-week, open-label study. J Diabetes Investig. 2016 Jan;7(1):100-8. doi: 10.1111/jdi.12361. Epub 2015 May 18. PMID 26816607
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study, F1J-JE-HMFY (Study HMFY), is an open-label, long-term extension study of double-blind placebo-controlled study F1J-JE-HMFX (Study HMFX) (NCT00552175).
Pre-assignment Details: Prior to start of extension study (HMFY), all participants in Study HMFX were re-randomized to duloxetine 40 or 60 mg regardless of the treatment they received in Study HMFX. Baseline values for the extension study HMFY represent those of 40- and 60-mg groups after re-randomization of participants.
Groups:
- Duloxetine 40 mg: Duloxetine 40 mg once daily (QD), orally (PO), 1 year
Period: Overall Study
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Started | 129 | 129
Completed | 99 | 92 (1 participant discontinued during taper phase, not during treatment phase.)
Not Completed | 30 | 37
Not completed — Lack of Efficacy | 1 | 2
Not completed — Adverse Event | 24 | 29
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Reason Not Specified | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 129 | 129 | 258
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (10.5) | 60.0 (9.6) | 60.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 22 | 62
  Male | 89 | 107 | 196
Race/Ethnicity, Customized [Number; unit: participants] — All participants were Japanese.
  participants | 129 | 129 | 258
Region of Enrollment [Number; unit: participants]
  Japan | 129 | 129 | 258
Duration of Diabetes [Number; unit: participants]
  Less Than 5 Years | 23 | 25 | 48
  5 to 10 Years | 27 | 23 | 50
  Greater Than or Equal to 10 Years | 76 | 79 | 155
  Unknown | 3 | 2 | 5
Type of Diabetes [Number; unit: participants] — Type I diabetes is insulin dependent diabetes. Type II diabetes is non-insulin dependent diabetes.
  participants
    Type I | 8 | 4 | 12
    Type II | 121 | 125 | 246
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 163.69 (9.04) | 165.12 (7.75) | 164.41 (8.44)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 63.91 (12.13) | 64.98 (11.57) | 64.45 (11.84)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meters squared (kg/m^2)] — Body mass index (BMI) is an estimate of body fat based on body weight divided by height squared (kg/m^2).
  kilograms/meters squared (kg/m^2) | 23.79 (3.77) | 23.77 (3.49) | 23.78 (3.62)
Duration of Diabetic Neuropathy [Mean (Standard Deviation); unit: years] | 3.91 (3.16) | 4.29 (3.91) | 4.10 (3.55)
Patient's Global Impressions of Improvement (PGI-I) Rate [Mean (Standard Deviation); unit: units on a scale] — A scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
  units on a scale | 3.0 (1.1) | 3.1 (1.1) | 3.1 (1.1)
Beck Depression Inventory - II (BDI-II) [Mean (Standard Deviation); unit: units on a scale] — A 21-item, participant-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a 4-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
  units on a scale | 6.1 (6.4) | 6.1 (6.4) | 6.1 (6.4)
Brief Pain Inventory (BPI) Interference [Mean (Standard Deviation); unit: units on a scale] — Self-reported scale measures interference of pain on function in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life. Scores range from 0 (does not interfere) to 10 (completely interferes). Average interference = self-reported scale measures interference of pain on average of 7 questions assessing interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life. Average Interference scores range from 0 (does not interfere) to 10 (completely interferes).
  units on a scale
    General Activity | 2.5 (2.4) | 2.7 (2.2) | 2.6 (2.3)
    Mood | 2.3 (2.3) | 2.4 (2.2) | 2.3 (2.2)
    Walking Ability | 2.2 (2.4) | 2.3 (2.1) | 2.3 (2.2)
    Normal Work | 2.3 (2.3) | 2.3 (2.2) | 2.3 (2.3)
    Relation to People | 1.6 (2.1) | 1.9 (2.1) | 1.8 (2.1)
    Sleep | 2.2 (2.3) | 2.5 (2.4) | 2.3 (2.4)
    Enjoyment of Life | 1.9 (2.1) | 2.1 (2.1) | 2.0 (2.1)
    Average Interference Score | 2.14 (2.09) | 2.32 (2.06) | 2.23 (2.07)
Brief Pain Inventory (BPI) - Pain Severity [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain, least pain, and worst pain experienced over the past 24 hours, and the pain right now. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale
    Worst Pain | 4.7 (2.0) | 4.9 (2.0) | 4.8 (2.0)
    Least Pain | 2.8 (2.0) | 3.1 (2.1) | 3.0 (2.0)
    Average Pain | 3.8 (1.9) | 4.0 (1.9) | 3.9 (1.9)
    Pain Right Now | 3.4 (2.1) | 3.6 (2.1) | 3.5 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: See the Reported Adverse Events section for details.
Time Frame: baseline through 1 year
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 129
participants
  Serious Adverse Events | 11 | 22
  Adverse Events | 126 | 121

2. Secondary Outcome: Patient Global Impression of Improvement (PGI-I) Scale at One Year Endpoint.
Description: A scale that measures the participant's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: 1 year
Population: Intention to treat (ITT) population - participants were analyzed according to the groups to which they were originally assigned, whether or not they completed the protocol.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale | 2.1 (0.9) | 2.1 (1.0)

3. Secondary Outcome: Change From Baseline to One Year Endpoint for Patient Global Impression of Improvement (PGI-I) Scale
Description: as for outcome 2
Time Frame: baseline, 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale | -0.9 (1.1) | -1.0 (1.1)

4. Secondary Outcome: Brief Pain Inventory (BPI) Severity Scores at One Year Endpoint
Description: A self-reported scale that measures the severity of pain. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). There are 4 questions assessing worst pain, least pain, and average pain in the past 24 hours, and the pain right now.
Time Frame: 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale
  Worst Pain | 2.4 (1.9) | 2.6 (2.0)
  Least Pain | 1.3 (1.5) | 1.5 (1.5)
  Average Pain | 1.8 (1.5) | 1.9 (1.6)
  Pain Right Now | 1.7 (1.6) | 1.7 (1.6)

5. Secondary Outcome: Change From Baseline to One Year Endpoint in Brief Pain Inventory (BPI) Severity Scores
Description: as for outcome 4
Time Frame: baseline, 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale
  Worst Pain | -2.2 (1.8) | -2.3 (1.9)
  Least Pain | -1.6 (1.6) | -1.6 (1.6)
  Average Pain | -2.1 (1.7) | -2.1 (1.6)
  Pain Right Now | -1.8 (1.7) | -1.8 (1.6)

6. Secondary Outcome: Brief Pain Inventory (BPI) Interference Scores at One Year Endpoint
Description: Self-reported scale measures interference of pain on function in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life. Scores range from 0 (does not interfere) to 10 (completely interferes). Average interference = self-reported scale measures interference of pain on average of 7 questions assessing interference of pain for general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life. Average interference scores range from 0 (does not interfere) to 10 (completely interferes).
Time Frame: 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale
  General Activities | 1.4 (1.7) | 1.4 (1.6)
  Mood | 1.2 (1.5) | 1.3 (1.6)
  Walking Ability | 1.4 (1.7) | 1.3 (1.5)
  Normal Work | 1.2 (1.7) | 1.3 (1.5)
  Relation to People | 1.0 (1.5) | 1.1 (1.4)
  Sleep | 1.2 (1.5) | 1.3 (1.6)
  Enjoyment of Life | 1.2 (1.6) | 1.3 (1.5)
  Average Score | 1.21 (1.52) | 1.28 (1.48)

7. Secondary Outcome: Change From Baseline to One Year Endpoint in Brief Pain Inventory (BPI) Interference Scores
Description: as for outcome 6
Time Frame: baseline, 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale
  General Activities | -1.1 (1.8) | -1.3 (1.8)
  Mood | -1.1 (1.8) | -1.0 (1.7)
  Walking Ability | -0.8 (1.8) | -1.0 (1.6)
  Normal Work | -1.0 (1.8) | -1.0 (1.6)
  Relation to People | -0.6 (1.6) | -0.7 (1.6)
  Sleep | -1.0 (2.1) | -1.1 (2.0)
  Enjoyment of Life | -0.8 (1.7) | -0.8 (1.5)
  Average Score | -0.93 (1.57) | -1.00 (1.48)

8. Secondary Outcome: Beck Depression Inventory-II (BDI-II) Total Score at One Year Endpoint
Description: A 21-item, participant-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a 4-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Time Frame: 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale | 6.3 (7.1) | 5.4 (5.8)

9. Secondary Outcome: Change From Baseline to One Year Endpoint in Beck Depression Inventory-II (BDI-II) Total Score
Description: as for outcome 8
Time Frame: baseline, 1 year
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Number analyzed (Participants) | 129 | 128
units on a scale | 0.2 (4.4) | -0.7 (3.7)

ADVERSE EVENTS:
Arm/Group | Duloxetine 40 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 11/129 | 22/129
Other Adverse Events (participants affected / at risk) | 126/129 | 121/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 40 mg (N=129) | Duloxetine 60 mg (N=129)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Infected epidermal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pyonephrosis (Infections and infestations) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vertebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine 40 mg (N=129) | Duloxetine 60 mg (N=129)
Diabetic retinopathy (Eye disorders) | 8 (8) | 3 (3)
Constipation (Gastrointestinal disorders) | 17 (19) | 17 (19)
Diarrhoea (Gastrointestinal disorders) | 9 (10) | 7 (7)
Nausea (Gastrointestinal disorders) | 14 (16) | 13 (15)
Stomach discomfort (Gastrointestinal disorders) | 4 (7) | 7 (7)
Vomiting (Gastrointestinal disorders) | 9 (11) | 10 (12)
Oedema peripheral (General disorders) | 7 (9) | 8 (8)
Thirst (General disorders) | 5 (5) | 8 (9)
Nasopharyngitis (Infections and infestations) | 36 (52) | 31 (39)
Pharyngitis (Infections and infestations) | 5 (6) | 11 (12)
Contusion (Injury, poisoning and procedural complications) | 10 (11) | 12 (20)
Alanine aminotransferase increased (Investigations) | 12 (12) | 13 (15)
Aspartate aminotransferase increased (Investigations) | 13 (13) | 12 (14)
Blood alkaline phosphatase increased (Investigations) | 6 (6) | 7 (8)
Blood creatine phosphokinase increased (Investigations) | 12 (13) | 12 (12)
Blood creatinine increased (Investigations) | 3 (4) | 8 (9)
Blood glucose decreased (Investigations) | 14 (22) | 8 (9)
Blood glucose increased (Investigations) | 14 (21) | 12 (14)
Blood lactate dehydrogenase increased (Investigations) | 7 (7) | 5 (5)
Blood potassium increased (Investigations) | 7 (8) | 7 (10)
Blood triglycerides increased (Investigations) | 9 (11) | 10 (10)
Blood urea increased (Investigations) | 7 (7) | 4 (4)
Blood uric acid increased (Investigations) | 6 (7) | 8 (8)
Blood urine present (Investigations) | 4 (4) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 10 (10) | 11 (11)
Glycosylated haemoglobin increased (Investigations) | 31 (32) | 29 (29)
Urine albumin/creatinine ratio increased (Investigations) | 10 (11) | 15 (15)
Weight increased (Investigations) | 12 (13) | 11 (11)
White blood cell count increased (Investigations) | 13 (16) | 8 (8)
Diabetes mellitus (Metabolism and nutrition disorders) | 12 (13) | 11 (11)
Hypoglycaemia (Metabolism and nutrition disorders) | 14 (34) | 11 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 9 (10)
Dizziness (Nervous system disorders) | 10 (12) | 8 (11)
Headache (Nervous system disorders) | 11 (31) | 9 (13)
Somnolence (Nervous system disorders) | 17 (17) | 18 (18)
Insomnia (Psychiatric disorders) | 11 (11) | 5 (5)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9 (14) | 3 (6)
Eczema (Skin and subcutaneous tissue disorders) | 8 (9) | 10 (14)
Hypertension (Vascular disorders) | 9 (12) | 8 (8)
Orthostatic hypotension (Vascular disorders) | 4 (4) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days